CLINICAL TRIAL: NCT05885802
Title: The Role of Sngception and Pain in Enhanced Recovery After Surgery (ERAS) for Spine Surgeries
Brief Title: Sngception and Pain in Spine Enhanced Recovery After Surgery (ERAS) Pathways
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 2022-09-009BC
Record Dates: First submitted 2023-05-16; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pain Postoperative
Keywords: enhanced recovery; ERAS; Spine surgery; pain; sngception; sng
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERAS group: Routine spine surgical patients receiving ERAS protocol that complies with current guidelines.
  Interventions: Other: No specific intervention other than routine anesthesia protocol

INTERVENTIONS:
Other: No specific intervention other than routine anesthesia protocol — No specific intervention other than routine anesthesia protocol

SUMMARY:
Enhanced recovery after surgery (ERAS) is a recognized, evidence-based and patient-centered clinical pathway that has an array of benefits. Minimally invasive techniques, a cyclopedic pain management plan and precise administration of anesthetics, which will render patients a rapid and comfortable recovery if executed correctly, followed by early mobilization and discharge.

Pain management practice is traveling through a paradigm shift as opioid crises arise in the western countries. Opioid-based pain control is being disarmed and replaced by multimodal analgesia (MMA) and becoming the mainstay strategy. Opioids are increasingly being reserved as rescue medications. MMA target different parts of the nociceptive pathway, preventing its wind-up during surgery. Decreased firing of the nociceptive neurons may be linked to lower postoperative pain scores or even the suppressing chronic pain incidence. In our ERAS pathway, we implement erector spinae plane block (ESPB) as the main analgesic firepower.

As postoperative pain decreases, an observed rising complaint is "sng", or soreness, in native Taiwanese in our ERAS spine patients. It is very different from the nociceptive "pain" we are familiar with. Patients avoid movements if it causes pain, but they tend to stretch or adjust postures if sngception dominates. The term "sngception" has been proposed in 2018 by Taiwanese scholars. It is believed to be a sense of acidosis, possibly within the muscles. Acidosis and associated pain are well documented, such as in muscle aches from exercise, cancer or diabetic ketoacidosis. The underlying mechanism is yet to be established but does not entirely overlap with nociception. There are numerous similarities of sngception in our patients and sngception:

1. a sensation different from nociception,
2. usual painkillers are ineffective, suggesting an alternative route of transmission,
3. relieved by movement,
4. inflammation and acidosis in the vicinity of surgical wound. In this study, we intended to characterize sngception by observing various perioperative factors, as well as the short- and long- term outcomes they bring. This will be done through a detailed sngception and pain trajectory analysis. Only when we know the main causative factor(s), we can design treatment plans toward guarding against sngception. This further improves the quality of postoperative recovery and safety as less opioids may be required as rescue medications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing routine ERAS protocol for spine surgeries
2. American Society of Anesthesiologists Physical Status (ASA-PS) I~III

Exclusion Criteria:

1. Communication issues that preclude proper preoperative counselling for ERAS and study design.
2. Active alcohol or drug addiction.
3. Pregnancy
4. Allergy to main anesthetics that preclude the use of routine ERAS anesthesia management.
5. Patient refusal to participate in study.
6. Emergent operations.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving routine ERAS management for spine surgeries. All patients will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative Sngception (Sng) | From enrollment to 1 year after surgery.
  Sng score evaluated by the numerical rating scale (NRS, score 0~10).
Postoperative Pain | From enrollment to 1 year after surgery.
  Pain score evaluated by the numerical rating scale (NRS, score 0~10).

SECONDARY OUTCOMES:
Morphine consumption | From enrollment to discharge, an average of 5 days.
  Postoperative morphine consumption converted to Morphine Sulfate Equivalents (MSE)

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei City, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin JH, Hung CH, Han DS, Chen ST, Lee CH, Sun WZ, Chen CC. Sensing acidosis: nociception or sngception? J Biomed Sci. 2018 Nov 29;25(1):85. doi: 10.1186/s12929-018-0486-5. PMID 30486810